CLINICAL TRIAL: NCT06251596
Title: What is the Impact of Frozen Embryo Transfer Protocol, on Endometrial Compaction
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0202-20-HYMC
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-02

CONDITIONS: IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ovulatory cycles: Patients with ovulatory cycles
- Patients with artificial cycles: Patients with artificial cycles

SUMMARY:
This study aims to evaluate endometrial thickness on the day of the frozen embryo transfer, compared to endometrial thickness on the last day of assessment of the endometrium before exposure to progesterone in respect to the protocols used for endometrial preparation

DETAILED DESCRIPTION:
247 FET cycles were included in the study. Records of all patients and their cryopreservation embryos were analyzed. Data collection included baseline parameters of age, BMI (kg/m2), type of infertility, parity, lifestyles, and cause of infertility, as well as treatment parameters, including number of embryos transferred, embryo quality and pregnancy outcomes.

To reflect the broad range of patients typically encountered in clinical practice, no inclusion/exclusion criteria were applied regarding baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Pregnancy

Ages: 20 Years to 44 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Females only
Study Population: 250 IVF patients undergoing the return of frozen embryos
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Endometrial compaction in each group. | 5 years
  Endometrial compaction in each group.

SECONDARY OUTCOMES:
Implantation and pregnancy rates in each group | 5 years
  Implantation and pregnancy rates in each group

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom Paz, PROF, Principal Investigator — Israel Hillel Yaffe medical center; Anna Turetzky Oved, Nurse, Study Chair — Israel Hillel Yaffe medical center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Heifa Region, Israel